CLINICAL TRIAL: NCT06030973
Title: Opinions of Healthcare Providers About a European Neuromodulation Register: an Online Survey
Brief Title: Opinions of Healthcare Providers About a European Neuromodulation Register
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moens Maarten (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, Principal Investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: PROLOGUE
Record Dates: First submitted 2023-08-26; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Registry; Neuromodulation; Survey

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare professionals involved in neuromodulation
  Interventions: Behavioral: Filling in an online survey

INTERVENTIONS:
Behavioral: Filling in an online survey — Professionals are asked to complete questions regarding 1) the degree of current participation in a registry, 2) the need for a European registry, 3) the items that should be collected and 4) access to the European registry.

SUMMARY:
The goal of this online survey is to gain further insights in the needs and burden for a European registry for neuromodulation, according to healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults who are involved in the management of chronic pain and more specifically in neuromodulation for pain (including but not limited to anesthesiologists, neurosurgeons, nurses).

Exclusion Criteria:

* Not involved in management of chronic pain through neuromodulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study male and female adults who are involved in the management of chronic pain and more specifically in neuromodulation for pain (including but not limited to anesthesiologists, neurosurgeons, nurses) will be eligible to complete the survey. The survey will be spread at the 3ʳᵈ Joint Congress of the INS European Chapters (e-INS 2023) in Hamburg from 31/8/2023 to 2/9/2023.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2023-09-02 (Estimated); Study Completion 2023-09-02 (Estimated)

PRIMARY OUTCOMES:
Healthcare providers their current degree of participation in a registry for neuromodulation. | Cross-sectional evaluation during 3th Joint Congress of the INS European Chapters (e-INS 2023) in Hamburg in August-September 2023.
  Degree of participation in a registry for neuromodulation (question).
Healthcare providers their need for a European registry. | Cross-sectional evaluation during 3th Joint Congress of the INS European Chapters (e-INS 2023) in Hamburg in August-September 2023.
  Underlying reasons on why a European registry is needed, or not needed (question).
Items that should be included in a registry for neuromodulation, according to healthcare providers. | Cross-sectional evaluation during 3th Joint Congress of the INS European Chapters (e-INS 2023) in Hamburg in August-September 2023.
  Items that should be collection within a registry, evaluated with a multiple choice question.
Access regulations to European registry for neuromodulation, according to healthcare providers. | Cross-sectional evaluation during 3th Joint Congress of the INS European Chapters (e-INS 2023) in Hamburg in August-September 2023.
  Access regulations, evaluated with a multiple choice question.

CONTACTS AND LOCATIONS:
Locations (1):
- Congres Center, Hamburg, Germany